CLINICAL TRIAL: NCT03374436
Title: Salivary Insulin Profiles Throughout the Day in Healthy Humans
Brief Title: Impact of Sprint Stair Climbing "Snacks" on Markers of Metabolism and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Mitacs (Industry); CoreHealth Technologies Inc. (Unknown)
Responsible Party: Principal Investigator, Jonathan Little, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: H17-01747
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Physical Activity; Diet Modification
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants complete three conditions in a repeated crossover design.
Masking Description: It is not possible to mask the exercise or diet interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-Carbohydrate Sedentary (Experimental): Participants will remain seated for 9 hours (except for using the restroom) while consuming a high-carbohydrate diet (3 meals)
  Interventions: Behavioral: High-Carbohydrate Sedentary
- High-Carbohydrate Active (Experimental): Participants will remain seated for 9 hours (except for using the restroom) while consuming a high-carbohydrate diet (3 meals) but will complete 8 stair climbing sprint "snacks" once per hour involving ascending 3 flights of stairs at a vigorous pace (~20 seconds each).
  Interventions: Behavioral: High-Carbohydrate Active
- Low-Carbohydrate Sedentary (Active Comparator): Participants will remain seated for 9 hours (except for using the restroom) while consuming a low-carbohydrate diet (3 meals)
  Interventions: Behavioral: Low-carbohydrate Sedentary

INTERVENTIONS:
Behavioral: High-Carbohydrate Sedentary — Three high-carbohydrate meals will be consumed (breakfast, lunch, and dinner) at ~3 hour intervals while participants remain in a seated position for the entire 9 hour intervention period.
  Arms: High-Carbohydrate Sedentary
Behavioral: High-Carbohydrate Active — Three high-carbohydrate meals will be consumed (breakfast, lunch, and dinner) at ~3 hour intervals while participants remain in a seated position for the entire 9 hour intervention period except that once every hour they will ascend three flights of stairs vigorously (stair climbing sprint "snack") for a total of 8 active breaks.
  Arms: High-Carbohydrate Active
Behavioral: Low-carbohydrate Sedentary — Three low-carbohydrate meals will be consumed (breakfast, lunch, and dinner) at ~3 hour intervals while participants remain in a seated position for the entire 9 hour intervention period. This condition will provide a condition where the blood glucose and insulin responses are relatively low and stable throughout the day.
  Arms: Low-Carbohydrate Sedentary

SUMMARY:
Prolonged sitting has been shown to impair metabolism and vascular function. The overall purpose of this study is to determine if breaking up prolonged (9 hours) of sitting with brief (~20 second) stair climbing exercise "snacks" can improve markers of metabolic control and vascular health in healthy young male participants and in males or females with overweight/obesity who are at risk of insulin resistance. An additional purpose is to determine if saliva insulin can be used as a valid indicator of blood insulin when measured throughout the day in sedentary and active conditions and when diets with different amounts of carbohydrates are consumed.

ELIGIBILITY:
Lean Group Inclusion Criteria:

Non-smoking

Lean Group Exclusion Criteria:

Diagnosed with diabetes or prediabetes (fasting blood sugar more than 6.0 mmol/l) or any other chronic condition that may impact glucose or insulin levels.

BMI is over 25 kg/m2 Take medications which may affect glucose and insulin levels Allergic to eggs. Smoker Competitive or serious endurance athlete.

Overweight/Obese Group Inclusion Criteria:

Elevated waist circumference (>102 cm for male and >88 cm for female)

Overweight/Obese Group Exclusion Criteria:

Diagnosed with diabetes (fasting blood sugar more than 7.0 mmol/l) Take medications which may affect glucose and insulin levels Allergic to eggs. Smoker Competitive or serious endurance athlete.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Plasma insulin area under the curve | Measured across 9 hours of each intervention day
  The plasma insulin concentration measured by enzyme-linked immunosorbent assay area under the curve will be measured using the trapezoidal rule.

SECONDARY OUTCOMES:
Saliva insulin area under the curve | Measured across 9 hours of each intervention day
  The saliva insulin concentration measured by enzyme-linked immunosorbent assay area under the curve will be measured using the trapezoidal rule.
Plasma glucose area under the curve | Measured across 9 hours of each intervention day
  The plasma glucose concentration measured by hexokinase method area under the curve will be measured using the trapezoidal rule.
Plasma triglyceride area under the curve | Measured across 9 hours of each intervention day
  The plasma triglyceride concentration measured by biochemical assay area under the curve will be measured using the trapezoidal rule.
Plasma non-esterified fatty acids area under the curve | Measured across 9 hours of each intervention day
  The plasma non-esterified fatty acid concentration measured by biochemical assay area under the curve will be measured using the trapezoidal rule.
Femoral artery flow-mediated dilation | Measured in the morning (time 0 hours) and afternoon (time 8.5 hours) each intervention day
  Flow-mediated dilation of femoral artery measured by vascular ultrasound
Cerebrovascular function | Measured in the morning (time 0.5 hours) and afternoon (time 6 hours) each intervention day
  Cerebrovascular function measured by transcranial doppler ultrasound
Cognitive function | Measured in the morning (time 0.5 hours) and afternoon (time 6 hours) each intervention day
  Cognitive function measured by Computerized Neurocognitive Assessment Software (CNS) Vital Signs test battery

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
We will share individual patient data (de-identified) with researchers upon request.

REFERENCES:
- [Derived] Rafiei H, Omidian K, Chang CR, Little JP. Saliva insulin tracks plasma insulin across the day following high-carbohydrate and low-carbohydrate meals. Appl Physiol Nutr Metab. 2023 Sep 1;48(9):700-709. doi: 10.1139/apnm-2023-0066. Epub 2023 Jun 1. PMID 37262929
- [Derived] Caldwell HG, Coombs GB, Rafiei H, Ainslie PN, Little JP. Hourly staircase sprinting exercise "snacks" improve femoral artery shear patterns but not flow-mediated dilation or cerebrovascular regulation: a pilot study. Appl Physiol Nutr Metab. 2021 May;46(5):521-529. doi: 10.1139/apnm-2020-0562. Epub 2020 Nov 26. PMID 33242251